CLINICAL TRIAL: NCT03582319
Title: Clinical and Radiographic Evaluation of Biodentine Versus Formocresol in Vital Pulpotomy of Primary Molars: (A Randomized Control Clinical Trial)
Brief Title: Clinical and Radiographic Evaluation of Biodentine Versus Formocresol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Adel Abdel Azeem Elbardissy, Associate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Abardissy
Record Dates: First submitted 2018-06-03; First posted 2018-07-11 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Pulp Disease, Dental
MeSH Terms: conditions — Dental Pulp Diseases | interventions — tricalcium silicate; formocresol

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, double blinded using split mouth technique.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biodentine (Experimental): Regenerative material for pulp therapy
  Interventions: Other: Biodentine
- Formocresol (Active Comparator): Fixative agent for pulp therapy
  Interventions: Other: Formocresol

INTERVENTIONS:
Other: Biodentine — Biodentine is mainly composed of tricalcium silicate, calcium carbonate and zirconium oxides while the liquid contains calcium chloride as the setting accelerator and water reducing agent
  Arms: Biodentine
Other: Formocresol — Formocresol is a devitalizing and fixing agent which was introduced to dentistry since 1904 with full concentration of Buckley's formula (19% formaldehyde, 35 % cresol, and 15 % glycerin in distilled water). A five times diluted formula of Buckley's formocresol was used in this study.
  Other Names: Tricresol formalin
  Arms: Formocresol

SUMMARY:
Aim of the study: To compare Formocresol and Biodentine clinically and radiographically when used for pulpotomy of primary molars Study Design : A randomized control clinical trial (split mouth and double blind) was conducted on 43 (4-6 years-old) children with decayed vital mandibular primary molars which were treated by pulpotomy using both medicaments . All treated teeth were followed for one year (at 3, 6, 9 and 12 months clinically and at 6 and 9 radiographically).

DETAILED DESCRIPTION:
Study design Randomized clinical trial, double blinded using split mouth technique. Study setting This study was carried out in Pediatric Dentistry Department-Faculty of Dentistry-Cairo University- Egypt.

Patients

Patients recruited for this study were selected according to the following criteria:

* Healthy children between 4 and 6 years of age with two matched bilateral deep carious primary mandibular first or second molars.
* No evident clinical symptoms of pulpal necrosis or pulp degeneration such as pain on percussion, spontaneous pain, history of swelling or presence of sinus tract.
* No pathologic or physiologic mobility.
* No radiographic evidence of internal and external resorption, pulp stone, and interradicular or periapical lesions (Preoperative radiograph).
* The remaining tooth structure would be restorable with a stainless steel crown.
* Bleeding time after amputation of the coronal pulp tissue was within normal limits (5 minutes).

Sample size calculation using sealedenvelop.com, (30) the online sample calculator, sample size was calculated assuming the null hypothesis that biodentine and formocresol have an average success rate of 95,99 % and 87.8 % respectively (26, 31,32,33). Thus planning a binary outcome non inferiority trial with a difference of 8.19 %, then 76 primary molars (38 per group) are required to be 90% sure that the upper limit of a one-sided 95% confidence interval will exclude a difference in favor of the standard group of more than 10% (34).

With an estimation of 10% annual dropout, sample size was set to 86 primary molars (43 per group) (35). Forty three children with the matching criteria of patient selection were included in this study.

Research Ethics Committee approval was obtained from Faculty of Dentistry Cairo University. Detailed treatment plan and procedures were explained to the parents and informed written consent s were obtained before practical work.

Randomization Using 4 times folded papers in which one of the tested materials was written (43 paper for each material) contained in a closed white envelops (43 envelop in each one folded paper of each tested materials were placed), the selected two matched bilateral deep carious primary mandibular molars were randomly allocated to one of the tested materials.

When guardians agreed for their child to participate in the trial, an envelope was drowned and patient personal data was written on it. At the time of treatment of the first tooth in each patient, one of the folded papers was taken from the envelope and the type of the dressing material was recorded. Trial participant and outcome assessors were blinded to the type of materials used in each tooth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between 4 and 6 years of age with two matched bilateral deep carious primary mandibular first or second molars.
* No evident clinical symptoms of pulpal necrosis or pulp degeneration such as pain on percussion, spontaneous pain, history of swelling or presence of sinus tract.
* No pathologic or physiologic mobility.
* No radiographic evidence of internal and external resorption, pulp stone, and interradicular or periapical lesions (Preoperative radiograph).
* The remaining tooth structure would be restorable with a stainless steel crown.
* Bleeding time after amputation of the coronal pulp tissue was within normal limits (5 minutes).

Exclusion Criteria:

* Bleeding time after amputation of the coronal pulp tissue exceed normal limits (5 minutes).

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2017-02-12 (Actual); Primary Completion 2018-01-20 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Assessing survival rate regarding absence of spontaneous pain over time. using a questionnaire. | 3,6,9 and12 months.
  measurement of survival rate regarding absence of spontaneous pain and assessing the change over time ( binary outcome measured by direct questioning to the patient.

SECONDARY OUTCOMES:
Assessing absence of abscess, fistula or pathologic mobility over time using visual and clinical examination. | 3, 6, 9 and 12 months.
  Absence of abscess, fistula or pathologic mobility ( binary outcome measured by visual and clinical examination).
Absence of periapical or inter-radicular radiolucency (binary outcome detected by periapical x-ray ). | 6 and 12 months.
  Absence of periapical or inter-radicular radiolucency (binary outcome detected by periapical x-ray ) with assessment of change over time.
Absence of external or internal root resorption(binary outcome detected by periapical x-ray ) . | 6 and 12 months
  Absence of external or internal root resorption(binary outcome detected by periapical x-ray ) with assessment of change over time.
Absence of calcific metamorphosis in the radicular pulp canal (binary outcome detected by periapical x-ray ) . | 6 and 12 months
  Absence of calcific metamorphosis in the radicular pulp canal (binary outcome detected by periapical x-ray ) with assessment of change over time.

CONTACTS AND LOCATIONS:
Locations (1):
- Adel Elbardissy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No